CLINICAL TRIAL: NCT03051958
Title: Internet-based Mindfulness and Exposure Treatment for Atopic Dermatitis: Randomized Controlled Trial
Brief Title: Internet-based Mindfulness and Exposure Treatment for Atopic Dermatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Erik Hedman, PhD, associate professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ICBT atopic dermatitis
Record Dates: First submitted 2017-01-23; First posted 2017-02-14 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internet mindfulness&exposure treatment (Experimental): A 12-week treatment where the main treatment components are mindfulness, exposure and response prevention, a form of cognitive behavior therapy. The treatment entails methods to increase acceptance and non-reactivity to aversive thoughts and emotions associated with AD. The treatment is delivered via the Internet and comprises 10 modules, each with a specific theme. Throughout treatment, the patient is given structured exercises to work with on a daily basis.
  Interventions: Behavioral: Internet mindfulness&exposure treatment
- Treatment as usual (Active Comparator): Participants receive information about moisturizer and anti-inflammatory lotion treatment which is treatment as usual.
  After 12 weeks, patients in this arm are crossed over to treatment.
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Behavioral: Internet mindfulness&exposure treatment — See description under "Arm".
  Other Names: I-MET
  Arms: Internet mindfulness&exposure treatment
Other: Treatment as usual — Written information about standard treatment for atopic dermatitis, that is information regarding how to use moisturizers and anti-inflammatory treatment such as Topical steroids.
  Arms: Treatment as usual

SUMMARY:
Atopic dermatitis (AD) is highly prevalent and leads to suffering for the individual, increased risk of depressive symptoms and anxiety, and high societal costs. A few psychological treatment have been tested for AD, but to our knowledge none of them have been built on recently developed methods for optimizing exposure treatment. In addition, access to psychological treatment is limited and there is a need for new methods that could be easily disseminated. One possible solution to this problem is to deliver psychological treatment via the Internet, which has been tested in more than 100 randomized trials with good results for other clinical disorders than AD. The aim of this study was to test the effects of Internet-delivered mindfulness and exposure treatment (I-MET) for AD in a randomized controlled trial. We hypothesized that I-MET would lead to larger reductions of AD symptoms as well as psychological symptoms compared to treatment as usual.

DETAILED DESCRIPTION:
Atopic dermatitis (AD), characterized by chronic itching and inflammation, is highly prevalent and leads to suffering for the individual, increased risk of depressive symptoms and anxiety, and high societal costs. Several behavioral factors are likely to play a role in the exacerbating AD symptoms over time, not least scratching, which may lead to rupture in the skin barrier and an increased risk of inflammation, which in turns increases AD symptoms. AD is also associated with avoidance behaviors that may have negative longer-term effects. With this in mind, psychological treatment based on exposure may be a logical method to achieve improvements. A few psychological treatments have been tested for AD, but to our knowledge none of them have been built on recently developed methods for optimizing exposure treatment. In a recently conducted pilot study we showed that exposure treatment, in combination with mindfulness training, can be associated with improvements for persons with AD. One challenge regarding psychological treatment is that accessibility is limited and there is a need for new methods that could be easily disseminated. One possible solution to this problem is to deliver psychological treatment via the Internet, which has been tested in more than 100 randomized trials with good results for other clinical disorders than AD. Internet-based treatment can be described as a form of online bibliotherapy where the individual is guided by a therapist who provides feedback on homework assignments. The aim of this study was to test the effects of Internet-delivered mindfulness and exposure treatment (I-MET) for AD in a randomized controlled trial. We hypothesized that I-MET would lead to larger reductions of AD symptoms as well perceived stress, sleep problems, depressive symptoms, general anxiety, and improved self-rated health, compared to treatment as usual.

CLARIFICATION REGARDING STUDY START DATE (remark made on March 15, 2021): This trial employed one informed consent which was completed before the provision of screening data for the purpose of assessing eligibility. The first date on which a participant provided informed consent and screening data was Nov 27, 2016. The first date a participant was included in the study, as based on the assessment of eligibility criteria in accordance with the study protocol, was March 29, 2017. The latter date is considered to be the study start date, in accordance with 81 FR 65022.

ELIGIBILITY:
Inclusion Criteria:

* Fulfills the diagnostic criteria for atopic dermatitis in accordance with Williams criteria 1994
* at the time of inclusion the eczema should be at least moderate according to The Patient Oriented Eczema Measure (POEM)
* Regular access to computer and internet connection
* If on antidepressant or regular sleep medication, the medication should be stable for at least one month prior to inclusion and the person should be willing to keep the medication stable throughout the study
* possibility to actively carry out the treatment (not go for longer journeys, do homework)
* good understanding of written and spoken Swedish

Exclusion Criteria:

* severe psychiatric illness (bipolar disorder, schizophrenia or other psychotic illness, substance, alcohol abuse, severe depression, suicide risk)
* difficulties with reading or writing
* ongoing treatment for cancer
* pregnancy
* other psychological treatment that i ongoing or recently terminated
* stronger anxiety-reducing medication such as benzodiazepines
* treatment with antibiotics that is ongoing or has been terminated less than one month prior to inclusion
* Psoriasis
* UV-light treatment that is ongoing or has been terminated less than one month prior to inclusion
* oral treatment for eczema that is ongoing or has been terminated less than two month prior to inclusion

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2017-03-29 (Actual); Primary Completion 2019-06-28 (Actual); Study Completion 2019-06-28 (Actual)

PRIMARY OUTCOMES:
Patient-Oriented Eczema Measure (POEM) | baseline, week 1, week 2, week 3, week 4, week 5, week 6, week 7, week 8, week 9, week 10, week 11, post-treatment (12 weeks) , 6 month follow-up, 12 month follow-up
  Change in POEM at post-treatment and 6 and 12 month follow-ups compared to baseline

SECONDARY OUTCOMES:
Visual analogue scale itch (VAS-itch) | baseline, week 1, week 2, week 3, week 4, week 5, week 6, week 7, week 8, week 9, week 10, week 11, post-treatment (12 weeks), weekly during treatment, 6 month follow-up, 12 month follow-up
  Change in VAS-scratch at post-treatment and 6 and 12 month follow-ups compared to baseline
Visual analogue scale scratch (VAS-scratch) | baseline, week 1, week 2, week 3, week 4, week 5, week 6, week 7, week 8, week 9, week 10, week 11, post-treatment (12 weeks), 6 month follow-up, 12 month follow-up
  Change in VAS-scratch at post-treatment and 6 and 12 month follow-ups compared to baseline
Visual analogue scale sleep (VAS-sleep) | baseline, week 1, week 2, week 3, week 4, week 5, week 6, week 7, week 8, week 9, week 10, week 11, post-treatment (12 weeks), 6 month follow-up, 12 month follow-up
  Change in VAS-sleep at post-treatment and 6 and 12 month follow-ups compared to baseline
Dermatology Quality of Life Index (DLQI) | baseline, post-treatment (12 weeks), 6 month follow-up, 12 month follow-up
  Change in DLQI at post-treatment and 6 and 12 month follow-ups compared to baseline
Beck Anxiety Inventory (BAI) | baseline, post-treatment (12 weeks), 6 month follow-up, 12 month follow-up
  Change in BAI at post-treatment and 6 and 12 month follow-ups compared to baseline
Patient Health Questionnaire-9 (PHQ-9) | baseline, post-treatment (12 weeks), 6 month follow-up, 12 month follow-up
  Change in PHQ-9 at post-treatment and 6 and 12 month follow-ups compared to baseline
Perceived stress scale (PSS) | baseline, post-treatment (12 weeks), 6 month follow-up, 12 month follow-up
  Change in PSS at post-treatment and 6 and 12 month follow-ups compared to baseline
5-dimensions itch scale (5-D itch scale) | baseline, post-treatment (12 weeks), 6 month follow-up, 12 month follow-up
  Change in 5-D itch scale at post-treatment and 6 and 12 month follow-ups compared to baseline
Insomnia Severity Index (ISI) | baseline, post-treatment (12 weeks), 6 month follow-up, 12 month follow-up
  Change in ISI at post-treatment and 6 and 12 month follow-ups compared to baseline
Self-Rated Health (SRH-5) | baseline, post-treatment (12 weeks), 6 month follow-up, 12 month follow-up
  Change in SRH-5 at post-treatment and 6 and 12 month follow-ups compared to baseline
Brunnsviken Brief Quality of life scale (BBQ) | baseline, post-treatment (12 weeks), 6 month follow-up, 12 month follow-up
  Change in BBQ at post-treatment and 6 and 12 month follow-ups compared to baseline
EuroQoL-5 Dimension Questionnaire (EQ-5D) | baseline, post-treatment (12 weeks), 6 month follow-up, 12 month follow-up
  Change in EQ5D at post-treatment and 6 and 12 month follow-ups compared to baseline
The Trimbos and Institute for Medical Technology Assessment Questionnaire on Costs Associated with Psychiatric Illness (TIC-P) | baseline, post-treatment (12 weeks), 6 month follow-up, 12 month follow-up
  Change in TIC-P at post-treatment and 6 and 12 month follow-ups compared to baseline

OTHER OUTCOMES:
Client Satisfaction Questionnaire (CSQ-8) | Post-treatment (12)
  Mean and standard deviations will be presented
Alcohol Disorders Identification Test (AUDIT) | Baseline
  This measure is used only as a mean for gathering data regarding inclusion/exclusion criteria
Drug Use Disorders Identification Test (DUDIT) | Baseline
  This measure is used only as a mean for gathering data regarding inclusion/exclusion criteria
Mediators using: Pain Reactivity Scale, Psychological Inflexibility in Pain Scale, Five Facets of Mindfulness- non reactivity scale, visual analogue scales for (itch, scratching and insomnia), and use of antiinflammatory skin creme | baseline, week 1, week 2, week 3, week 4, week 5, week 6, week 7, week 8, week 9, week 10, week 11, post-treatment (12 weeks)
  Change in mediators from baseline to post-treatment (12 weeks) will be correlated with change in the primary outcome during the same time period

CONTACTS AND LOCATIONS:
Overall Officials: Erik Hedman, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No
Karolinska Institutet requires that a formal assessment if the data can be made public must be conducted before publishing individual level data

REFERENCES:
- [Derived] Hedman-Lagerlof E, Fust J, Axelsson E, Bonnert M, Lalouni M, Molander O, Agrell P, Bergman A, Lindefors N, Bradley M. Internet-Delivered Cognitive Behavior Therapy for Atopic Dermatitis: A Randomized Clinical Trial. JAMA Dermatol. 2021 Jul 1;157(7):796-804. doi: 10.1001/jamadermatol.2021.1450. PMID 34009282